CLINICAL TRIAL: NCT03088254
Title: A Multi-center, Randomized, Double-blind, Parellel Phase III Clinical Trial to Evaluate the Efficacy and Safety of Triple Therapy of Telmisartan/Amlodipine/Rosuvastatin in Patients With Dyslipidemia and Hypertension
Brief Title: Study to Evaluate the Efficacy and Safety of Telmisartan/Amlodipine/Rosuvastatin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jeil Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: J-TAROS-RCT
Record Dates: First submitted 2017-03-08; First posted 2017-03-23 (Actual); Last update posted 2018-07-06 (Actual); Status verified 2018-03

CONDITIONS: Dyslipidemia With Hypertension
MeSH Terms: interventions — Telmisartan; Amlodipine; Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I (Experimental): Treatment of Telmisartan 80 mg, Amodipine 10 mg, Rosuvastatin 20 mg for 8 weeks
  Interventions: Drug: Group I (Telmisartan 80 mg, Amlodipine 10 mg, Rosuvastatin 20 mg)
- Group II (Active Comparator): Treatment of Telmisartan 80 mg, Amodipine 10 mg, Rosuvastatin placebo for 8 weeks
  Interventions: Drug: Group II (Telmisartan 80 mg, Amodipine 10 mg, Rosuvastatin placebo)
- Group III (Active Comparator): Treatment of Telmisartan 80 mg, Amodipine placebo, Rosuvastatin 20 mg for 8 weeks
  Interventions: Drug: Group III (Telmisartan 80 mg, Amlodipine placebo, Rosuvastatin 20 mg)

INTERVENTIONS:
Drug: Group I (Telmisartan 80 mg, Amlodipine 10 mg, Rosuvastatin 20 mg) — Twinstar(80/10 mg) and Rosuvastatin 20 mg for 8 weeks
  Arms: Group I
Drug: Group II (Telmisartan 80 mg, Amodipine 10 mg, Rosuvastatin placebo) — Twinstar(80/10 mg) and Rosuvastatin placebo for 8 weeks
  Arms: Group II
Drug: Group III (Telmisartan 80 mg, Amlodipine placebo, Rosuvastatin 20 mg) — Twinstar placebo, Amlodipine 10 mg and Rosuvastatin 20 mg for 8 weeks
  Arms: Group III

SUMMARY:
To evaluate efficacy and safety of co-administrated temisartan/amlodipine and rosuvastatin in subjects with dyslipidemia with hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Dyslipidemia with hypertesion
* msSBP < 180 mmHg
* msDBP < 110 mmHg
* LDL-C ≤ 250 mg/dL
* Triglycerides < 400 mg/dL

Exclusion Criteria:

* At Visit 3, BP difference SBP ≥20mmHg or DBP ≥10mmHg
* CK normal range ≥ 2 times
* Uncontrolled primary hypothyroidism(TSH normal range ≥ 1.5 times)
* AST or ALT ≥ 2 times
* Uncontrolled diabetes mellitus (HbA1c≥9%)
* CLcr < 30 mL/min/1.73m^2
* K > 5.5 mEq/L
* Other exclusion applied

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2016-09-20 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-12-04 (Actual)

PRIMARY OUTCOMES:
change of LDL-C | baseline and 8 weeks
change of msSBP | baseline and 8 weeks

CONTACTS AND LOCATIONS:
Locations (12):
- South Korea (12):
  - Chungnam National University Hospital, Daejeon
  - Chonnam National University Hospital, Gwangju
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Gachon University Gil Medical Center, Incheon
  - Inje University Haeundae Paik Hospital, Pusan
  - Ewha Womans University Mokdong Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - KyungHee University Hospital at Gangdong, Seoul
  - Seoul National University Hospital, Seoul
  - SoonChunHyang University Hospital, Seoul, Seoul
  - The Catholic University of Korea Seoul St. Mary's Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hong SJ, Jeong HS, Cho JM, Chang K, Pyun WB, Ahn Y, Hyon MS, Kang WC, Lee JH, Kim HS. Efficacy and Safety of Triple Therapy With Telmisartan, Amlodipine, and Rosuvastatin in Patients With Dyslipidemia and Hypertension: The Jeil Telmisartan, Amlodipine, and Rosuvastatin Randomized Clinical Trial. Clin Ther. 2019 Feb;41(2):233-248.e9. doi: 10.1016/j.clinthera.2018.12.008. Epub 2019 Jan 18. PMID 30665829